CLINICAL TRIAL: NCT01851733
Title: A Pilot Study of Using MRI-Guided Laser Heat Ablation to Induce Disruption of the Peritumoral Blood Brain Barrier to Enhance Delivery and Efficacy of Doxorubicin in the Treatment of Recurrent Glioblastoma Multiforme
Brief Title: MRI-Guided Laser Surgery and Doxorubicin Hydrochloride in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201305148
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Doxorubicin; Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm B: (MLA, doxorubicin hydrochloride at 6-8 weeks) (Experimental): * Patients undergo MLA (MRI-guided laser heat ablation). A subset of patients will have a biopsy at time of MLA.
  * Beginning 6-8 weeks later, patients receive doxorubicin hydrochloride 20 mg/m2 intravenously (IV) over 5 minutes once weekly for 6 weeks.
  * Biomarker blood draws will be drawn at different time points.
  * DSC-MRI: no more than 2 weeks prior to MLA, within approximately 3 days after MLA, 2/4/6 weeks after MLA, 10 weeks after MLA only if 6-week scan shows prolonged disruption of the blood brain barrier, 14 weeks after MLA only if week 10 MRI shows contined blood brain barrier disruption, and every 8 weeks until disease progression (these scans do not have to be DSC-MRI)
  Interventions: Device: MRI-guided Laser Heat Ablation (MLA); Drug: Doxorubicin; Other: Blood draw - dendritic cells; Device: Dynamic Susceptibility Contrast Magnetic Resonance Imaging
- Arm C: (MLA, doxorubicin hydrochloride at 72 hours) (Experimental): * Patients undergo MLA (MRI-guided laser heat ablation).
  * Beginning within 72 hours later, patients receive doxorubicin hydrochloride 20 mg/m2 IV over 5 minutes once weekly for 6 weeks.
    * DSC-MRI: no more than 2 weeks prior to MLA, within approximately 3 days after MLA, 2/4/6 weeks after MLA, 10 weeks after MLA only if 6-week scan shows prolonged disruption of the blood brain barrier, 14 weeks after MLA only if week 10 MRI shows contined blood brain barrier disruption, and every 8 weeks until disease progression (these scans do not have to be DSC-MRI)
  Interventions: Device: MRI-guided Laser Heat Ablation (MLA); Drug: Doxorubicin; Device: Dynamic Susceptibility Contrast Magnetic Resonance Imaging

INTERVENTIONS:
Device: MRI-guided Laser Heat Ablation (MLA)
Drug: Doxorubicin
  Other Names: Adriamycin®
Other: Blood draw - dendritic cells — The second 10 patients enrolled to Arm B:
  * before MLA (up to 3 days before)
  * 2 weeks after MLA
  * 4 weeks after MLA
  * every 2 weeks thereafter for up to 3 months after biopsy (provided there is no significant chemotherapy induced cytopenia)
  Arms: Arm B: (MLA, doxorubicin hydrochloride at 6-8 weeks)
Device: Dynamic Susceptibility Contrast Magnetic Resonance Imaging
  Other Names: DSC-MRI

SUMMARY:
This pilot clinical trial studies magnetic resonance imaging (MRI)-guided laser surgery (MLA) and doxorubicin hydrochloride in treating patients with recurrent glioblastoma multiforme. The blood brain barrier (BBB) is a separation of circulating blood from the tissue of the central nervous system, preventing substances in the blood from entering the brain. MLA disrupts the BBB around the tumor which may allow cancer-killing substances to be carried directly to the tumor and the surrounding area. Using MLA prior to chemotherapy may result in a greater concentration of drug in the tumor to kill the cancer cells while limiting side effects.

DETAILED DESCRIPTION:
Evaluate imaging techniques (MRI) and blood tests (biomarkers) to help figure out the best time for chemotherapy to be initiated after the blood brain barrier is disrupted, as it is immediately following a procedure like MRI-guided laser ablation (MLA-Monteris Neuroblate).

ELIGIBILITY:
Inclusion Criteria - Arms B and C:

* Histologically confirmed GBM; rare GBM variants, secondary GBM, and suspected secondary GBM are allowed.
* Unequivocal evidence of tumor progression by magnetic resonance imaging (MRI) scan.
* There must be an interval of at least 12 weeks from the completion of radiotherapy to study registration except if there is unequivocal evidence for tumor recurrence per RANO criteria. When the interval is less than 12 weeks from the completion of radiotherapy, the use of PET scan is allowed to differentiate between unequivocal evidence of tumor recurrence and pseudoprogression.
* Candidate for MLA based on size, location, and shape of the recurrent tumor as determined by the performing neurosurgeon
* At least 18 years of age.
* Karnofsky performance status ≥ 60%.
* Scheduled for MRI-guided Laser Ablation (MLA).
* Normal left ventricular ejection fraction on MUGA or echocardiogram within the past 1 year prior to registration for patients with history of congestive heart failure and/or coronary disease requiring medications other than aspirin, or known prior exposure to anthracycline chemotherapy.
* Adequate bone marrow and hepatic function as defined below (must be within 7 days of MLA):

  * Absolute neutrophil count (ANC) ≥ 1500/mcl (G-CSF is allowed)
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9 (pRBC transfusion +/- ESA are allowed)
  * ALT ≤ 3 x ULN
  * AST ≤ 3 x ULN
  * ALP ≤ 3 x ULN. If ALP is > 3 x ULN, GGT must be checked and be ≤ 3 x ULN.
  * Bilirubin ≤ 2 x ULN
* At the time of registration, patient must have recovered from the toxic effects of prior therapy to no more than grade 1 toxicity.
* At the time of registration, patient must be at least 2 weeks from prior vincristine, 3 weeks from prior procarbazine, and 4 weeks from other prior cytotoxic chemotherapy.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria - Arms B and C:

* Prior treatment with doxorubicin and/or bevacizumab.
* Prior treatment with Gliadel wafer is allowed if it has been at least 3 months from placement.
* Previous treatment with complete cumulative doses of daunorubicin, idarubicin, and/or other anthracyclines and anthracenediones that is equivalent to a total dose of 240 mg/m2 doxorubicin.
* More than 2 prior relapses.
* Currently receiving any other investigational agents that are intended as treatments of GBM.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to doxorubicin or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recent heart attack within the previous 12 months or severe heart problems, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Premenopausal women must have a negative serum pregnancy test within 14 days of study entry.
* Inability to undergo MRI due to personal and medical reasons.
* Known history of HIV or autoimmune diseases requiring immunosuppressant drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Ktrans from DSC-MRI | 6 weeks
  Using a 2 compartment model to calculate a the vascular transfer constant (Ktrans) which will provide a quantitative measure of blood brain barrier leakage
Peritumoral permeability scores, measured by DSC-MRI and serum biomarkers | 6 weeks
  Pearson correlation coefficient (r) will be determined for each biomarker and Ktrans value. A minimum r=0.5 is required for inclusion for further analysis and will be used as a peritumoral permeability score. This score will then be correlated with the patient outcome data to determine whether it has a predictive value.
6-month PFS (rate) | 6 months
  Assessed using RANO Response criteria. A log-rank test will be used to compare 6-PFS of Arm B and of Arm C to historical controls.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Date began MLA treatment to date of death from any cause. A log-rank test will be used to compare OS of Arm B and of Arm C to historical controls.
Quality of Life | 2 years
  Using Karnofsky performance status and the mini-mental state evaluation to assess patient overall response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Chheda, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leuthardt EC, Duan C, Kim MJ, Campian JL, Kim AH, Miller-Thomas MM, Shimony JS, Tran DD. Hyperthermic Laser Ablation of Recurrent Glioblastoma Leads to Temporary Disruption of the Peritumoral Blood Brain Barrier. PLoS One. 2016 Feb 24;11(2):e0148613. doi: 10.1371/journal.pone.0148613. eCollection 2016. PMID 26910903
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu